CLINICAL TRIAL: NCT07237815
Title: Exploring the Quiet Quitting Phenomenon in Physiotherapy - A Cross Sectional Study
Brief Title: The Quiet Quitting Phenomenon Among Physiotherapists
Acronym: Quiet Quitting
Status: Completed | Type: Observational
Sponsor: Regione del Veneto - AULSS n. 7 Pedemontana (Other)
Responsible Party: Principal Investigator, Eleonora Lazzaretti, Principal Investigator - PT, MSC, Adjunct Professor at the University of Padua, Regione del Veneto - AULSS n. 7 Pedemontana
Other Study IDs: 699 CET
Record Dates: First submitted 2025-08-19; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Quiet Quitting
Keywords: job satisfaction; lack of initiative; lack of motivation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: Questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire consists of three sections, structured as follows: The introductory section is dedicated to verifying compliance with the inclusion criteria, which include: age of 18 years or older, and the provision of informed consent to participate in the study. Following these three initial questions, four additional items are included to collect basic demographic and occupational information from participants: gender, age group, years of work experience, level of education, and primary work setting. The second section comprises the items from the Job Satisfaction Survey (JSS).
  This assessment tool has already been validated in its Italian version through the study conducted by Platania and collaborators. The third section of the questionnaire is dedicated to the Quiet Quitting Scale (QQS), which includes nine items grouped into three latent factors: • detachment (4 items) • lack of initiative (3 items) • lack of motivation (2 items)

SUMMARY:
The COVID-19 pandemic has profoundly impacted all aspects of human life. Health work professsions have faced the risk of infection, adverse working conditions, physical and verbal violence, disparities in workload and payment, limitations to attend social activities, and disruption in work-life balance for a long time. The inadequacy of attempts to solve the issues caused them to change their work attitudes and behaviours, highlighting the ongoing need for a healthier work-life balance. In this context, a new trend known as 'quiet quitting' has emerged. This concept represents a notable workplace phenomenon, especially in settings with high demands and intense workloads. Quiet quitting refers to a situation where employees perform only the minimum requirements of their job description, refraining from any extra effort, innovation, or contribution beyond the bare minimum. Employees who begin the process of quiet quitting may exhibit behaviours such as leaving the workplace early, arriving at work late, refusing to engage in work outside working hours, demonstrating a lack of interest in assisting coworkers, and resisting going above and beyond minimum job duties. Individuals who are in the process of quiet quitting are emotionally detached from their jobs. This is a factor that profoundly impacts healthcare services. Although the quiet quitting process, which results in reduced productivity, increased employee turnover and decreased work quality, as well as negative consequences for patient safety and satisfaction, helps employees avoid burnout, it can jeopardize their career advancement. Furthermore, lower levels of job satisfaction appear to be associated with higher levels of quiet quitting among employees.

DETAILED DESCRIPTION:
Health workers are essential to the functioning of health systems; expanding health care coverage and attaining the right to the highest possible level of health are based on the availability, accessibility, acceptance, and quality of health care. Policymakers must take the necessary steps to improve health care quality by considering gender, family, profession, and age group differences in line with technological, scientific, and social developments. Additionally, the investigators need to remember the factors that reduce organizational commitment, job satisfaction, productivity, and motivation. Acting in the international cooperation framework will contribute to greater harmony between societies.

The identified study design is an observational study without the use of drugs or medical devices. The study involved the use of a questionnaire specifically structured for this research, divided into three distinct sections. The first section is aimed at collecting demographic and professional data from participants, as well as verifying compliance with the inclusion criteria. The second section includes the 36 items of the Job Satisfaction Survey (JSS), translated into Italian. Finally, the third section consists of the 9 items of the Quiet Quitting Scale, also translated into Italian. Sampling will follow a non-probability approach, using convenience sampling. Participants will be recruited through the dissemination of a questionnaire created with Google Forms. Recruitment will occur via the institutional channels (newsletter/website) of the Professional Board of Physiotherapists of Belluno- Treviso-Vicenza-Verona and the Italian Association of Physiotherapists (AIFI) - Veneto section, subject to prior authorization, along with a request for voluntary participation. Individuals who respond to the questionnaire, provide informed consent, and meet the inclusion criteria will be enrolled in the study. All participants will be included and the questionnaire will be administered at a single time point (T0); no follow-up is planned. Reading and accepting the study information sheet-after reviewing the data processing information and providing informed consent-will be considered an essential condition for questionnaire administration, as outlined in the information notice. The consent form and information sheet will be integrated into the Google Forms format, and only after selecting "Yes, I Consent" for both fields (data processing and informed consent) on the first page will the respondent be granted access to the actual questionnaire. It will not be possible to trace the participant's email address or IP address. To achieve the targeted sample size, the questionnaire will be disseminated through the institutional channels of the Professional Board of Physiotherapists of Belluno-Treviso-Vicenza-Verona and the Italian Association of Physiotherapists (AIFI) - Veneto section, subject to prior authorization. Participation by physiotherapists will be voluntary. The communication will include the purpose of the survey, instructions for completing and submitting the questionnaire, and will consist of:

* A brief description of the study
* The information and informed consent form
* The information form regarding personal data processing
* Contact details of the study promoter for any additional information or clarifications
* A link to access the questionnaire Upon completion, by clicking "submit," respondents will send their responses to the electronic platform managed by the three project investigators. Thanks to a specific feature of Google Forms, each submission will be identified solely by the date and time of submission; it will not be possible to trace the participant's email address or IP address. In the absence of a randomized sample, the estimation of sample size is not considered binding. The study size will therefore be determined by the total number of participants who complete the questionnaire. However, although not binding, the following statistical guidelines are provided: with a 95% confidence level and an acceptable margin of error of 0.20, the goal is to estimate the mean score of the outcomes in the target population. The literature reports a standard deviation of 0.987, which will be adopted as a preliminary estimate of the standard deviation in this sample. Based on this information, a sample size of 94 participants is recommended to estimate the mean score of the outcomes. Means and standard deviations (medians and percentiles) will be calculated for continuous variables. For categorical variables, frequencies and proportions will be calculated. The association between the outcome and the variables of interest will be analyzed within each stratum of potential confounding factors (age, gender, years of experience). Scale scores between groups of interest (e.g., hospital vs. primary care) may be compared using appropriate statistical tests. The extent and nature of missing data will be assessed. In cases where a respondent has omitted a high number of responses, the entire questionnaire will be excluded. For small amounts of missing data, the missing values will be replaced by the median of the corresponding variable. Due to the use of convenience sampling, it is acknowledged that the sample may not be representative. Respondents with incomplete data will be excluded, and potential exclusion of outliers will also be considered.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists
* Aged 18 years or older
* Both genders

Exclusion Criteria:

* Presence of mental or physical conditions affecting the ability to understand or complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapist who work in the Veneto region (Italy) in all settings.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2025-10-23 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Quiet quitting phenomenon | baseline
  1. Quiet quitting phenomenon This study aims to investigate and explore the phenomenon of 'quiet quitting' within the healthcare rehabilitation sector, with a specific focus on physiotherapy personnel employed in hospital settings.
  The Quiet Quitting Scale (QQS) was administered in the third section. It is an instrument developed by Galanis et al. (2023a) to assess the phenomenon of quiet quitting. The scale consists of nine items organized into three factors: detachment (4 items), lack of initiative (3 items), and lack of motivation (2 items). Items are rated on a 5-point Likert scale (1 = strongly disagree; 5 = strongly agree).
  Interpretation of the mean score is straightforward: a value above 2.06 is used as a cut-off to indicate the presence of behaviors and attitudes associated with quiet quitting among professionals. Regarding the instrument's quality, the QQS was selected for its sound psychometric properties.

SECONDARY OUTCOMES:
Job satisfaction | baseline
  The secondary research question is addressed through the Job Satisfaction Survey (JSS). The Job Satisfaction Survey (JSS) was administered. This scale, developed by Spector (1985), measures job satisfaction. It consists of 36 items divided into nine dimensions: pay, promotion, supervision, benefits, contingent rewards, operating procedures, coworkers, nature of work, and communication. Each item is rated on a 6-point Likert scale (1 = strongly disagree; 6 = strongly agree).
  Interpretation of the mean score is structured across three levels, designed to clearly distinguish the degree of perceived job satisfaction among professionals:
  A score equal to or greater than 4 indicates job satisfaction.
  A score equal to or less than 3 reflects job dissatisfaction.
  Intermediate values between these two extremes are considered to express indifference or ambivalence toward one's work.
  To ensure the reliability of the results, the Italian version of the scale validated was used.

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS 7 Pedemontana, Bassano del Grappa, Vicenza, Italy

IPD SHARING:
Plan to Share IPD: No
IPD must be submitted to local Ethical Committee